CLINICAL TRIAL: NCT06869109
Title: Serum CXCL10 and CRP Levels in Patients with Acne Vulgaris in Correlation with Disease Severity
Acronym: CXCL10
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Essam, physician assiut university student hospital, Assiut University
Other Study IDs: role of CXCL10 and CRP in acne
Record Dates: First submitted 2025-03-04; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris; cxcl10; crp
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- mild acne group: mild disease severity
  Interventions: Diagnostic Test: serum cxcl10; Diagnostic Test: serum crp
- moderate acne group: moderate disease severity
  Interventions: Diagnostic Test: serum cxcl10; Diagnostic Test: serum crp
- severe acne group: severe disease severity
  Interventions: Diagnostic Test: serum cxcl10; Diagnostic Test: serum crp
- control group: healthy people
  Interventions: Diagnostic Test: serum cxcl10; Diagnostic Test: serum crp

INTERVENTIONS:
Diagnostic Test: serum cxcl10 — serum blood sample to measure the cxcl10
Diagnostic Test: serum crp — blood sample to measure crp

SUMMARY:
the correlations between CXCL10 levels, CRP, and acne severity scores (e.g., Global Acne Grading System) suggest that CXCL10 could serve as a biomarker of inflammation and acne severity. Understanding the relationship between CXCL10, CRP, and acne severity may offer insights into novel therapeutic strategies targeting inflammatory pathways in acne.

DETAILED DESCRIPTION:
Cross-sectional Observational Study. using 4 groups a 3 of different acne severity and controle one . the serum cxcl10 and crp will measured in each patient to correlate with disease severity

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 12-40 years diagnosed with acne vulgaris.
2. Both genders included.
3. Patients with mild, moderate, or severe acne severity as determined by a validated scoring system (e.g., Global Acne Grading System).
4. Patients not on systemic acne treatment (e.g., isotretinoin or antibiotics) or anti-inflammatory drugs.

Exclusion Criteria:

1. Patients with autoimmune diseases, systemic illnesses, acute infection or any other chronic inflammatory conditions that may affect CRP or CXCL10 levels.
2. Pregnant or lactating individuals.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: the patients with acne with different severity
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Correlation of CXCL10 and CRP levels with acne severity (GAG score). | within one year after the result
  compare the result of serum cxcl10 and crp with disease severity

SECONDARY OUTCOMES:
Identify thresholds of CXCL10 and CRP for predicting moderate/severe acne | within one year after the result
  the least result to identify the group
Explore potential differences based on sex or age groups | within one year of the result
  the effect of age and sex on the result

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Samir, prof, Study Director — Assiut University; Ahmed Shawky, prof, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abdelrazik YT, Ali FM, Salek MS, Finlay AY. Clinical experience and psychometric properties of the Cardiff Acne Disability Index (CADI). Br J Dermatol. 2021 Oct;185(4):711-724. doi: 10.1111/bjd.20391. Epub 2021 Jul 22. PMID 33864247
- [Background] Alsulaimani H, Kokandi A, Khawandanh S, Hamad R. Severity of Acne Vulgaris: Comparison of Two Assessment Methods. Clin Cosmet Investig Dermatol. 2020 Sep 28;13:711-716. doi: 10.2147/CCID.S266320. eCollection 2020. PMID 33061511
- [Background] Stańkowska A, Bergler-Czop B, Brzezińska-Wcisło L. Interleukins-6, -8 and -12p40 and C-reactive protein levels in patients with acne vulgaris with various severityof skin changes. Dermatology Review/Przegląd Dermatologiczny. 2020;107(4):308-22
- [Background] Yang CC, Huang YT, Yu CH, Wu MC, Hsu CC, Chen W. Inflammatory facial acne during uncomplicated pregnancy and post-partum in adult women: a preliminary hospital-based prospective observational study of 35 cases from Taiwan. J Eur Acad Dermatol Venereol. 2016 Oct;30(10):1787-1789. doi: 10.1111/jdv.13667. Epub 2016 Apr 22. PMID 27102946
- [Background] Kutlu O, Karadag AS, Unal E, Kelekci KH, Yalcinkaya Iyidal A, Topaloglu Demir F, Aksoy B, Colgecen E, Tosun M, Emre S, Tatliparmak A, Demirseren DD, Kaya Ozden H, Ozturk M, Ozlu E, Chen W. Acne in pregnancy: A prospective multicenter, cross-sectional study of 295 patients in Turkey. Int J Dermatol. 2020 Sep;59(9):1098-1105. doi: 10.1111/ijd.14999. Epub 2020 Jun 20. PMID 32562263
- [Background] Ansar W, Ghosh S, Ansar W, Ghosh S. Inflammation and inflammatory diseases, markers, and mediators: role of CRP in some inflammatory diseases. Biology of C reactive protein in health and disease. 2016:67-107
- [Background] Castell JV, Gomez-Lechon MJ, David M, Fabra R, Trullenque R, Heinrich PC. Acute-phase response of human hepatocytes: regulation of acute-phase protein synthesis by interleukin-6. Hepatology. 1990 Nov;12(5):1179-86. doi: 10.1002/hep.1840120517. PMID 1699862
- [Background] Yu H, Zhang B, Zhan Y, Yi Y, Jiang Q, Zhang Q, Wu Y, Wu M. Neutrophil extracellular trap-related mechanisms in acne vulgaris inspire a novel treatment strategy with adipose-derived stem cells. Sci Rep. 2024 Jan 17;14(1):1521. doi: 10.1038/s41598-024-51931-w. PMID 38233540
- [Background] Bowe WP, Logan AC. Clinical implications of lipid peroxidation in acne vulgaris: old wine in new bottles. Lipids Health Dis. 2010 Dec 9;9:141. doi: 10.1186/1476-511X-9-141. PMID 21143923
- [Background] Jin Z, Song Y, He L. A review of skin immune processes in acne. Front Immunol. 2023 Dec 15;14:1324930. doi: 10.3389/fimmu.2023.1324930. eCollection 2023. PMID 38193084
- [Background] Liang J, Chen Y, Wang Z, Wang Y, Mu S, Zhang D, Wang Z, Zeng W. Exploring the association between rosacea and acne by integrated bioinformatics analysis. Sci Rep. 2024 Feb 6;14(1):3065. doi: 10.1038/s41598-024-53453-x. PMID 38321132
- [Background] Williams HC, Dellavalle RP, Garner S. Acne vulgaris. Lancet. 2012 Jan 28;379(9813):361-72. doi: 10.1016/S0140-6736(11)60321-8. Epub 2011 Aug 29. PMID 21880356